CLINICAL TRIAL: NCT02745574
Title: Prevention of Post-laparoscopic Shoulder and Upper Abdominal Pain: A Randomized Controlled Trial.
Brief Title: Randomized Controlled Trail for Post Laparoscopic Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Principal Investigator, vghtpe user, YJ Chen, MD, PhD, deaprtment of Obstetrics and Gynecology, Taipei Veterans General Hospital, Taiwan
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 2013-04-038B
Record Dates: First submitted 2014-09-01; First posted 2016-04-20 (Estimated); Last update posted 2016-04-20 (Estimated); Status verified 2016-04

CONDITIONS: Shoulder Pain
Keywords: should and upper abdominal pain, post-laparoscopy
MeSH Terms: conditions — Shoulder Pain; Abdominal Pain | interventions — Saline Solution; Infusions, Parenteral

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Combined maneuver (Experimental): Combined maneuver: the upper part of the abdominal cavity was evenly and bilaterally filled with the 0.9% normal saline in the amount of 500 cc. We will leave the fluid in the abdominal cavity. Then, a pulmonary recruitment maneuver consisting of five manual pulmonary inflations was performed with a maximum pressure of 60 cm dihydrogen monoxide (H2O). The anesthesiologist held the fifth positive pressure inflation for approximately 5 seconds.
  Interventions: Procedure: Combined maneuver
- Intraperitoneal infusion (Experimental): the upper part of the abdominal cavity was evenly and bilaterally filled with the 0.9% normal saline in the amount of 500 cc. We will leave the fluid in the abdominal cavity.
  Interventions: Procedure: Intraperitoneal infusion
- Control group (No Intervention): CO2 was removed by passive exsufflation through the port site.

INTERVENTIONS:
Procedure: Combined maneuver — Combined maneuver (Intraperitoneal normal saline infusion and Pulmonary recruitment maneuver): the upper part of the abdominal cavity was evenly and bilaterally filled with the 0.9% normal saline in the amount of 500 cc. We will leave the 0.9% normal saline fluid in the abdominal cavity. Then, a pulmonary recruitment maneuver consisting of five manual pulmonary inflations was performed with a maximum pressure of 60 cm H2O. The anesthesiologist held the fifth positive pressure inflation for approximately 5 seconds.
  Other Names: 0.9% normal saline and manual pulmonary inflation
  Arms: Combined maneuver
Procedure: Intraperitoneal infusion — the upper part of the abdominal cavity was evenly and bilaterally filled with the 0.9% normal saline in the amount of 500 cc. We will leave the 0.9% normal saline fluid in the abdominal cavity.
  Other Names: 0.9% normal saline
  Arms: Intraperitoneal infusion

SUMMARY:
Laparoscopic surgery is becoming a major procedure, owing to smaller incisions, shorter hospitalizations, and less post-operative pain as compared with traditional laparotomies. However, there is marked interindividual variability of post-operative shoulder-tip pain following laparoscopic surgery. The incidence of shoulder pain varies from 35% to 80% and ranges from mild to severe. In some cases, it has been reported to last more than 72 hours after surgery.

The hypothesis of post-operative shoulder-tip pain is that carbon dioxide induced phrenic nerve irritation causes referred pain to C4. Therefore, we should try to do is that if we could reduce carbon dioxide retention in the pelvic cavity.

This clinical controlled trial is tried to find out the practical and clinical maneuver to reduce post-operative should-tip pain following laparoscopic surgery.

DETAILED DESCRIPTION:
All the patients will receive laparoscopic surgery using carbon dioxide (CO2 ) gas as distension medium. At the end of the surgery, in the control group C, CO2 was removed by passive exsufflation through the port site. In the intervention group A, at the end of the surgery, the upper part of the abdominal cavity was evenly and bilaterally filled with the 0.9% normal saline in the amount of 500 cc. We will leave the fluid in the abdominal cavity. Then, patients will be placed in the Trendelenburg position (30 degrees), and a pulmonary recruitment maneuver consisting of five manual pulmonary inflations was performed with a maximum pressure of 60 cm H2O. The anesthesiologists held the fifth positive pressure inflation for approximately 5 seconds. During these maneuvers, the surgeon was instructed to ensure that the trocar sleeve valve was fully open to allow the CO2 gas to escape.

In the intervention group B, at the end of the surgery, the upper part of the abdominal cavity was evenly and bilaterally filled with the 0.9% normal saline in the amount of 500 cc. We will leave the fluid in the abdominal cavity.

Patients will be asked to fill out questionnaires up to 48 hours to determine the frequency and severity of their shoulder and upper abdominal pain. The scores will be assessed 12, 24, 48 hours after surgery using a visual analogue scale( VAS) from 0 ( no pain) to 10 ( worst possible pain).

ELIGIBILITY:
Inclusion Criteria:

* Patients receive benign gynaecological laparoscopic surgery.
* American Society of Anesthesiologists (ASA) physical status of patient:

classification I-II

Exclusion Criteria:

* The procedure will be required to conversion to laparotomy.
* Any cardio-vascular diseases.

Ages: 20 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2013-04; Primary Completion 2017-01 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Change from baseline pain score of should and upper abdominal pain at 12 hours after surgery | Baseline and 12 hours after surgery
  The main objective of this trial is to assess the efficacy of clinical maneuver to reduce shoulder and upper abdominal pain. Thus the primary outcome measure of this trial is the severity and frequency of their should and upper abdominal pain.
  The pain score is based on the visual analogue scale in which patients record the intensity of their pain 12 hours after surgery. VAS consists of a subjective evaluation of the pain on a scale of 10 in which 0 is no pain and 10 the most severe pain.
Change from baseline pain score of should and upper abdominal pain at 24 hours after surgery | Baseline and 24 hours after surgery
  The main objective of this trial is to assess the efficacy of clinical maneuver to reduce shoulder and upper abdominal pain. Thus the primary outcome measure of this trial is the severity and frequency of their should and upper abdominal pain.
  The pain score is based on the visual analogue scale in which patients record the intensity of their pain 24 hours after surgery. VAS consists of a subjective evaluation of the pain on a scale of 10 in which 0 is no pain and 10 the most severe pain.
Change from baseline pain score of should and upper abdominal pain at 48 hours after surgery | Baseline and 48 hours after surgery
  The main objective of this trial is to assess the efficacy of clinical maneuver to reduce shoulder and upper abdominal pain. Thus the primary outcome measure of this trial is the severity and frequency of their should and upper abdominal pain.
  The pain score is based on the visual analogue scale in which patients record the intensity of their pain 48 hours after surgery. VAS consists of a subjective evaluation of the pain on a scale of 10 in which 0 is no pain and 10 the most severe pain.

SECONDARY OUTCOMES:
Change from baseline of Nause, vomiting and abdominal distention rate at 48 hours after surgery | Baseline and 48 hours after surgery
  Secondary outcome measures included the occurrence of nausea or vomiting and abdominal distention.

CONTACTS AND LOCATIONS:
Overall Officials: Yi Jen Chen, M.D., Ph.D., Study Chair — Taipei Veterans General Hospital, Taipei; Hsiao Wen Tsai, M.D., Principal Investigator — Taipei Veterans General Hostipal, Taipei
Locations (1):
- Taipei Veterans General Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Phelps P, Cakmakkaya OS, Apfel CC, Radke OC. A simple clinical maneuver to reduce laparoscopy-induced shoulder pain: a randomized controlled trial. Obstet Gynecol. 2008 May;111(5):1155-60. doi: 10.1097/AOG.0b013e31816e34b4. PMID 18448749
- [Result] Esmat ME, Elsebae MM, Nasr MM, Elsebaie SB. Combined low pressure pneumoperitoneum and intraperitoneal infusion of normal saline for reducing shoulder tip pain following laparoscopic cholecystectomy. World J Surg. 2006 Nov;30(11):1969-73. doi: 10.1007/s00268-005-0752-z. PMID 17043939